CLINICAL TRIAL: NCT05752994
Title: Effect of Multisensory Environment Room on Behavior in Children With Autism Spectrum Disorder
Brief Title: Multisensory Environment Room in Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sivaporn Vongpipatana, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2023/12
Record Dates: First submitted 2023-02-10; First posted 2023-03-03 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home program group (Active Comparator): The guardians will receive the education about autistic spectrum disorder and home program training.
  Interventions: Other: Home program
- Multisensory room group (Experimental): The guardians in this group will receiver the educational program the same as the home program group plus the training in multisensory room.
  Interventions: Other: Training in the multisensory room environment

INTERVENTIONS:
Other: Training in the multisensory room environment — The children will start with the swing follow with the scheduled activities and tabletop activity. The session will end in the relaxation room such as bubble tube, fiberoptic cascade, fiberoptic carpet and aurora projector bundle while the therapist has the interactive communication with children
  Arms: Multisensory room group
Other: Home program — Home program
  Arms: Home program group

SUMMARY:
To investigate the effect of multisensory environment room on behavior in children with autism spectrum disorder age 3-5 years old. The children will be randomized into 2 groups: the experimental and the control group. The control group will be educated about the autistic and hoe program training. The intervention group will got the same educational program as the control group plus training in multisensory room environment once a week for 10 weeks. The outcome measurement was done as the before intervention, at the 5th and 10th week.

DETAILED DESCRIPTION:
This project is a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* the children who was diagnosed with autism according to DSM-5
* age 3-5 years old
* has the severity mild-to-moderate and severe according to childhood autism rating scale, 2nd edition

Exclusion Criteria:

* The guardians deny to enroll into the study.
* blindness, deafness
* got the treatment of r-TMS less than 1 year

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Vineland Adaptive Behavior Scales-Third Edition (VABS-III) | baseline, change from baseline at 5 weeks, change from baseline at 10 weeks
  To measure communication, interpersonal skill and relationship of the children with autistm spectrum and other people in scales; 2 = often, 1= sometimes and 0= never. The minimum score is o. The max score in receptive domain is 78. The max score of expressive domain is 98. The max score of written domain is 76. The max score of personal domain is 110. The max score of domestic domain is 60. The max score of community domain is 116. The interpersonal relationships domain max score is 86. The max score of play and leisure domain is 72. The max score of copling skill domain is 66. The max score of gross motor domain is 86. The max score of fine motor domain is 68. The max score of maladaptive behavior domain is 88.

SECONDARY OUTCOMES:
Parent Stress Index 4th Edition: Short Form [PSI-4-SF] | baseline, change from baseline at 5 weeks, change from baseline at 10 weeks
  To measure stress in guardians with children with autism

CONTACTS AND LOCATIONS:
Overall Officials: Sivaporn Vongpipatana, MD., Principal Investigator — Department of Rehabilitation Medicine, Faculty of Medicine Ramathibodi Hospital Mahidol University
Locations (2):
- Thailand (2):
  - Chakri Naruebodindra Medical Institute, Bangkok, Changwat Samut Prakan
  - Faculty of Medicine Ramathibodi Hospital Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
The individual information of the subject will be concealed. The collected information will be shared for analysis.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The study protocol will be share among the researcher team to make a plan for data gathering and run the project. The statistical analytic plan and analytic code will be share among the data collector, statistician and primary investigator. The clinical study report will be share among the researcher team. The informed consent will be saved with the primary investigator.
Access Criteria: only among the researcher team

REFERENCES:
- [Background] Marco EJ, Hinkley LB, Hill SS, Nagarajan SS. Sensory processing in autism: a review of neurophysiologic findings. Pediatr Res. 2011 May;69(5 Pt 2):48R-54R. doi: 10.1203/PDR.0b013e3182130c54. PMID 21289533
- [Background] Shea N, Payne E, Russo N. Brief Report: Social Functioning Predicts Externalizing Problem Behaviors in Autism Spectrum Disorder. J Autism Dev Disord. 2018 Jun;48(6):2237-2242. doi: 10.1007/s10803-017-3459-8. PMID 29423607
- [Background] Sanchez A, Millan-Calenti JC, Lorenzo-Lopez L, Maseda A. Multisensory stimulation for people with dementia: a review of the literature. Am J Alzheimers Dis Other Demen. 2013 Feb;28(1):7-14. doi: 10.1177/1533317512466693. Epub 2012 Dec 7. PMID 23221029
- [Background] Unwin KL, Powell G, Jones CR. The use of Multi-Sensory Environments with autistic children: Exploring the effect of having control of sensory changes. Autism. 2022 Aug;26(6):1379-1394. doi: 10.1177/13623613211050176. Epub 2021 Oct 24. PMID 34693744
- [Background] Basadonne I, Cristofolini M, Mucchi I, Recla F, Bentenuto A, Zanella N. Working on Cognitive Functions in a Fully Digitalized Multisensory Interactive Room: A New Approach for Intervention in Autism Spectrum Disorders. Brain Sci. 2021 Nov 3;11(11):1459. doi: 10.3390/brainsci11111459. PMID 34827458
- [Background] Novakovic N, Milovancevic MP, Dejanovic SD, Aleksic B. Effects of Snoezelen-Multisensory environment on CARS scale in adolescents and adults with autism spectrum disorder. Res Dev Disabil. 2019 Jun;89:51-58. doi: 10.1016/j.ridd.2019.03.007. Epub 2019 Mar 29. PMID 30933867
- [Background] Staples KL, MacDonald M, Zimmer C. Assessment of motor behavior among children and adolescents with autism spectrum disorder. International Review of Research in Developmental Disabilities. 42: Elsevier; 2012. p. 179-214.
- [Background] Srikosai Soontaree, Moanchai Patcharee, Kamfou Chadaporn, Taweewattanaprecha Siriwan, Saipanish Ratana. ความ ตรง และ ความ เชื่อถือ ได้ ของ ดัชนี ชี้ วัด ความเครียด ผู้ ปกครอง ของ เด็ก อายุ 1เดือน ถึง 12 ปี. Journal of Mental Health of Thailand. 2020;28(1):56-71.
- [Background] Pajareya K, Sutchritpongsa S, Kongkasuwan R. DIR/Floortime® Parent Training Intervention for Children with Developmental Disabilities: a Randomized Controlled Trial. Siriraj Medical Journal. 2019;71(5):331- 38.
- [Background] American Psychiatric Association. The American Psychiatric Association's 2013 Annual Meeting. 2013. Contract No.: Abstract NR12-5
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, 5th ed.2014.
- See also: about the diagnosis of autism — https://www.psychiatry.org/psychiatrists/practice/dsm